CLINICAL TRIAL: NCT01545336
Title: A Double-blind, Placebo-controlled Phase II Study of Anastrozole in Patients With Pulmonary Arterial Hypertension
Brief Title: Anastrozole in Patients With Pulmonary Arterial Hypertension
Acronym: AIPH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 815035
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Anastrozole; Sugars; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anastrozole (Experimental): 1 mg tablet by mouth once daily for 3 months
  Interventions: Drug: Anastrozole
- Placebo (Placebo Comparator): Placebo tablet by mouth once daily for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anastrozole — 1 mg tablet to be taken 1 time daily
  Other Names: Arimidex
  Arms: Anastrozole
Drug: Placebo — 1 mg tablet to be taken 1 time daily
  Other Names: Sugar pill manufactured to mimic Anastrozole 1 mg tablet
  Arms: Placebo

SUMMARY:
The main purpose of this clinical trial is to study the safety and efficacy of anastrozole in adults diagnosed with pulmonary arterial hypertension (PAH). The study will evaluate how well the drug is tolerated. The study will also evaluate if anastrozole effects estradiol (E2) hormone levels, a sex hormone, and improves the function of the lower right chamber of the heart (right ventricle).

ELIGIBILITY:
Inclusion Criteria:

* Previous documentation of mean pulmonary artery pressure > 25 mm Hg with a pulmonary capillary wedge pressure (or left ventricular end-diastolic pressure) < 16 mm Hg and PVR > 3 WU at any time before study entry.
* Diagnosis of PAH which is idiopathic, heritable, drug- or toxin-induced, or associated with connective tissue disease, congenital heart disease, portal hypertension, or HIV infection.
* Most recent pulmonary function tests with FEV1/FVC >50% AND either a) total lung capacity > 70% predicted or b) total lung capacity between 60% and 70% predicted with no more than mild interstitial lung disease on computerized tomography scan of the chest
* Ability to perform six minute walk testing without limitations in musculoskeletal function or coordination.
* If female, post-menopausal state, defined as:
* > 50 years old AND
* a) have not menstruated during the preceding 12 months OR
* b) have follicle-stimulating hormone (FSH) levels (> 40 IU/L) OR
* < 50 years and FSH (> 40 IU/L) OR
* having had a bilateral oophorectomy
* Informed consent

Exclusion Criteria:

* Treatment with estrogen or anti-hormone therapy (tamoxifen, fulvestrant, etc.)
* WHO Class IV functional status
* History of breast cancer
* Clinically significant untreated sleep apnea
* Left-sided valvular disease (more than moderate mitral valve stenosis or insufficiency or aortic stenosis or insufficiency), pulmonary artery or valve stenosis, or ejection fraction < 45% on echocardiography
* Initiation of PAH therapy (prostacyclin analogues, endothelin-1 receptor antagonists, phosphodiesterase-5 inhibitors) within three months of enrollment; the dose must be stable for at least 3 months prior to Baseline Visit
* Hormone therapy
* Hospitalized or acutely ill
* Renal failure (creatinine > 2.0)
* Child-Pugh Class C cirrhosis
* Current or recent (< 6 months) chronic heavy alcohol consumption
* Current use of another investigational drug (non-FDA approved) for PAH
* Enrollment in a clinical trial within one month of screening
* Age < 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-10; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Kawut, MD, MS, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Pennsylvania - Penn Presbyterian, Philadelphia, Pennsylvania
  - University of Pennsylvania - Perelman Center, Philadelphia, Pennsylvania
  - Brown University - Rhode Island Hospital, Providence, Rhode Island

REFERENCES:
- [Result] Kawut SM, Archer-Chicko CL, DeMichele A, Fritz JS, Klinger JR, Ky B, Palevsky HI, Palmisciano AJ, Patel M, Pinder D, Propert KJ, Smith KA, Stanczyk F, Tracy R, Vaidya A, Whittenhall ME, Ventetuolo CE. Anastrozole in Pulmonary Arterial Hypertension. A Randomized, Double-Blind, Placebo-controlled Trial. Am J Respir Crit Care Med. 2017 Feb 1;195(3):360-368. doi: 10.1164/rccm.201605-1024OC. PMID 27602993

RESULTS

PARTICIPANT FLOW:
Groups:
- Anastrozole: Anastrozole 1 mg tablet by mouth once daily for 3 months
- Placebo: Placebo 1 mg tablet by mouth once daily for 3 months
Period: Overall Study
Arm/Group | Anastrozole | Placebo
Started | 12 | 6
Completed | 12 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anastrozole | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (13) | 59 (10) | 60.06 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 2 | 9
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 6 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 8 | 6 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 6 | 18
Six minute walk distance [Mean (Standard Deviation); unit: meters] | 336 (119) | 378 (161) | 350 (131)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Estradiol (E2) Level
Time Frame: Baseline, 3 months
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 12 | 6
% change from baseline | -40 [-61 to -26] | -4 [-14 to 4]

2. Primary Outcome: Tricuspid Annular Plane Systolic Excursion (TAPSE)
Time Frame: Baseline, 3 months
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 12 | 6
% change from baseline | 7 [0 to 28] | 10 [-6 to 33]

3. Secondary Outcome: Six Minute Walk Distance
Time Frame: Baseline, 3 months
Measure: Median (Inter-Quartile Range); unit: % change from baseline
Arm/Group | Anastrozole | Placebo
Number analyzed (Participants) | 12 | 6
% change from baseline | 8 [2 to 17] | -2 [-7 to 1]

ADVERSE EVENTS:
Time Frame: Adverse event data collected from Screening through 3 months
Arm/Group | Anastrozole | Placebo
Serious Adverse Events (participants affected / at risk) | 2/12 | 0/6
Other Adverse Events (participants affected / at risk) | 4/12 | 2/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=12) | Placebo (N=6)
Hemorrhoid: lower gastrointestinal bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anastrozole (N=12) | Placebo (N=6)
Myalgias (General disorders) | 4 (4) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fever (General disorders) | 2 (2) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (General disorders) | 1 (1) | 1 (1)
Confusion (General disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (General disorders) | 1 (1) | 2 (2)
Insomnia (General disorders) | 1 (1) | 0 (0)
Jaw pain (General disorders) | 1 (1) | 1 (1)
Oral thrush (General disorders) | 1 (1) | 0 (0)
Side cramps (General disorders) | 1 (1) | 0 (0)
Sinus congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight loss (General disorders) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 0 (0) | 1 (1)
Lightheadedness (General disorders) | 0 (0) | 1 (1)
Night sweats (General disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Presyncope (General disorders) | 0 (0) | 1 (1)
Worsening Raynaud's disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* Small sample size
* No changes in echo parameters
* Unclear mechanism for impact on 6MWD

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No